CLINICAL TRIAL: NCT01265498
Title: The Farnesoid X Receptor (FXR) Ligand Obeticholic Acid in Nonalcoholic Steatohepatitis (NASH) Treatment (FLINT) Trial
Brief Title: The Farnesoid X Receptor (FXR) Ligand Obeticholic Acid in NASH Treatment Trial(FLINT)
Acronym: FLINT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NASH-FLINT (IND); U01DK061730 (NIH)
Record Dates: First submitted 2010-12-21; First posted 2010-12-23 (Estimated); Results first posted 2015-08-21 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2015-07

CONDITIONS: Nonalcoholic Fatty Liver Disease (NAFLD); Nonalcoholic Steatohepatitis (NASH)
Keywords: Farnesoid X Receptor; FXR; Nonalcoholic fatty liver disease; Nonalcoholic steatohepatitis; NAFLD; NASH; obeticholic acid
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — obeticholic acid; farnesoid X-activated receptor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Obeticholic acid (Active Comparator): obeticholic acid
  Interventions: Drug: obeticholic acid
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: obeticholic acid — 25 mg daily for 72 weeks
  Other Names: farnesoid X receptor (FXR) ligand obeticholic acid (OCA)
  Arms: Obeticholic acid
Drug: placebo — placebo capsule, 25 mg daily for 72 weeks
  Other Names: Placebo for obeticholic acid
  Arms: Placebo

SUMMARY:
Administration of the farnesoid X receptor (FXR) ligand obeticholic acid (OCA) for 72 weeks to subjects with biopsy evidence of nonalcoholic steatohepatitis (NASH) will result in improvement in their liver disease as measured by changes in the nonalcoholic fatty liver disease (NAFLD) activity score (NAS).

DETAILED DESCRIPTION:
To evaluate whether treatment with obeticholic acid, 25 mg daily for 72 weeks compared to treatment with placebo, improves the severity of nonalcoholic fatty liver disease (NAFLD) as determined from hepatic histology.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older as of the initial screening interview and provision of consent
* Histologic evidence of definite or probable nonalcoholic steatohepatitis (NASH) based upon a liver biopsy obtained no more than 90 days prior to randomization and a nonalcoholic fatty liver disease activity score (NAS) of 4 or greater with at least 1 in each component of the NAS score (steatosis scored 0-3, ballooning degeneration scored 0-2, and lobular inflammation scored 0-3).

Exclusion Criteria:

* Current or history of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to screening (significant alcohol consumption is defined as more than 20 grams per day in females and more than 30 grams per day in males, on average)
* Inability to reliably quantify alcohol consumption based upon local study physician judgment
* Use of drugs historically associated with nonalcoholic fatty liver disease (NAFLD) (amiodarone, methotrexate, systemic glucocorticoids, tetracyclines, tamoxifen, estrogens at doses greater than those used for hormone replacement, anabolic steroids, valproic acid, and other known hepatotoxins) for more than 2 weeks in the year prior to randomization
* Prior or planned (during the study period) bariatric surgery (eg, gastroplasty, roux-en-Y gastric bypass)
* Uncontrolled diabetes defined as Hemoglobin A1c 9.5% or higher within 60 days prior to enrollment
* Presence of cirrhosis on liver biopsy
* A platelet count below 100,000/mm3
* Clinical evidence of hepatic decompensation as defined by the presence of any of the following abnormalities:

  * Serum albumin less than 3.2 grams/deciliter (g/dL)
  * International Normalized Ratio(INR)greater than 1.3
  * Direct bilirubin greater than 1.3 milligrams per deciliter (mg/dL)
  * History of esophageal varices, ascites or hepatic encephalopathy
* Evidence of other forms of chronic liver disease:

  * Hepatitis B as defined by presence of hepatitis B surface antigen (HBsAg)
  * Hepatitis C as defined by presence of hepatitis C virus (HCV) ribonucleic acid (RNA) or positive hepatitis C antibody (anti-HCV)
  * Evidence of ongoing autoimmune liver disease as defined by compatible liver histology
  * Primary biliary cirrhosis as defined by the presence of at least 2 of these criteria (i) Biochemical evidence of cholestasis based mainly on alkaline phosphatase elevation (ii)Presence of anti-mitochondrial antibody (AMA) (iii)Histologic evidence of nonsuppurative destructive cholangitis and destruction of interlobular bile ducts
  * Primary sclerosing cholangitis
  * Wilson's disease as defined by ceruloplasmin below the limits of normal and compatible liver histology
  * Alpha-1-antitrypsin(A1AT) deficiency as defined by diagnostic features in liver histology (confirmed by alpha-1 antitrypsin level less than normal; exclusion at the discretion of the study physician)
  * History of hemochromatosis or iron overload as defined by presence of 3+ or 4+ stainable iron on liver biopsy
  * Drug-induced liver disease as defined on the basis of typical exposure and history
  * Known bile duct obstruction
  * Suspected or proven liver cancer
  * Any other type of liver disease other than nonalcoholic steatohepatitis (NASH)
* Serum alanine aminotransferase (ALT) greater than 300 units per liter (U/L)
* Serum creatinine of 2.0 mg/dL or greater
* Use of ursodeoxycholic acid (Ursodiol, Urso) within 90 days prior to enrollment
* Inability to safely obtain a liver biopsy
* History of biliary diversion
* Known positivity for Human Immunodeficiency Virus (HIV) infection
* Active, serious medical disease with likely life expectancy less than 5 years
* Active substance abuse including inhaled or injection drugs in the year prior to screening
* Pregnancy, planned pregnancy, potential for pregnancy and unwillingness to use effective birth control during the trial, breast feeding
* Participation in an investigational new drug (IND) trial in the 30 days before randomization
* Any other condition which, in the opinion of the investigator, would impede compliance or hinder completion of the study
* Failure to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2011-03; Primary Completion 2014-01 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Doo, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (9):
- United States (9):
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Indiana University, Indianapolis, Indiana
  - St. Louis University, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Virginia Commonwealth University, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Shen W, Middleton MS, Cunha GM, Delgado TI, Wolfson T, Gamst A, Fowler KJ, Alazraki A, Trout AT, Ohliger MA, Shah SN, Bashir MR, Kleiner DE, Loomba R, Neuschwander-Tetri BA, Sanyal AJ, Zhou J, Sirlin CB, Lavine JE. Changes in abdominal adipose tissue depots assessed by MRI correlate with hepatic histologic improvement in non-alcoholic steatohepatitis. J Hepatol. 2023 Feb;78(2):238-246. doi: 10.1016/j.jhep.2022.10.027. Epub 2022 Nov 8. PMID 36368598
- [Derived] Vilar-Gomez E, Gawrieh S, Liang T, McIntyre AD, Hegele RA, Chalasani N. Interrogation of selected genes influencing serum LDL-Cholesterol levels in patients with well characterized NAFLD. J Clin Lipidol. 2021 Mar-Apr;15(2):275-291. doi: 10.1016/j.jacl.2020.12.010. Epub 2020 Dec 27. PMID 33454241
- [Derived] Loomba R, Neuschwander-Tetri BA, Sanyal A, Chalasani N, Diehl AM, Terrault N, Kowdley K, Dasarathy S, Kleiner D, Behling C, Lavine J, Van Natta M, Middleton M, Tonascia J, Sirlin C; NASH Clinical Research Network. Multicenter Validation of Association Between Decline in MRI-PDFF and Histologic Response in NASH. Hepatology. 2020 Oct;72(4):1219-1229. doi: 10.1002/hep.31121. Epub 2020 Oct 9. PMID 31965579
- [Derived] Siddiqui MS, Van Natta ML, Connelly MA, Vuppalanchi R, Neuschwander-Tetri BA, Tonascia J, Guy C, Loomba R, Dasarathy S, Wattacheril J, Chalasani N, Sanyal AJ; NASH CRN. Impact of obeticholic acid on the lipoprotein profile in patients with non-alcoholic steatohepatitis. J Hepatol. 2020 Jan;72(1):25-33. doi: 10.1016/j.jhep.2019.10.006. Epub 2019 Oct 18. PMID 31634532
- [Derived] Chalasani N, Abdelmalek MF, Loomba R, Kowdley KV, McCullough AJ, Dasarathy S, Neuschwander-Tetri BA, Terrault N, Ferguson B, Shringarpure R, Shapiro D, Sanyal AJ. Relationship between three commonly used non-invasive fibrosis biomarkers and improvement in fibrosis stage in patients with non-alcoholic steatohepatitis. Liver Int. 2019 May;39(5):924-932. doi: 10.1111/liv.13974. Epub 2019 Feb 21. PMID 30253043
- [Derived] Hameed B, Terrault NA, Gill RM, Loomba R, Chalasani N, Hoofnagle JH, Van Natta ML; NASH CRN. Clinical and metabolic effects associated with weight changes and obeticholic acid in non-alcoholic steatohepatitis. Aliment Pharmacol Ther. 2018 Mar;47(5):645-656. doi: 10.1111/apt.14492. Epub 2018 Jan 14. PMID 29333665
- [Derived] Neuschwander-Tetri BA, Loomba R, Sanyal AJ, Lavine JE, Van Natta ML, Abdelmalek MF, Chalasani N, Dasarathy S, Diehl AM, Hameed B, Kowdley KV, McCullough A, Terrault N, Clark JM, Tonascia J, Brunt EM, Kleiner DE, Doo E; NASH Clinical Research Network. Farnesoid X nuclear receptor ligand obeticholic acid for non-cirrhotic, non-alcoholic steatohepatitis (FLINT): a multicentre, randomised, placebo-controlled trial. Lancet. 2015 Mar 14;385(9972):956-65. doi: 10.1016/S0140-6736(14)61933-4. Epub 2014 Nov 7. PMID 25468160
- See also: Nonalcoholic Steatohepatitis Clinical Research Network — https://jhuccs1.us/nash/default.asp
- See also: The National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) — http://www2.niddk.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Obeticholic Acid | Placebo
Started | 141 | 142
Both Baseline and Week 72 Biopsy | 102 | 98
Completed | 110 | 109
Not Completed | 31 | 33
Not completed — Protocol modified to eliminate wk72 bx | 31 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Obeticholic Acid | Placebo | Total
Number analyzed (Participants) | 141 | 142 | 283
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (11) | 51 (12) | 51 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 89 | 187
  Male | 43 | 53 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 21 | 43
  Not Hispanic or Latino | 119 | 121 | 240
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 6 | 10 | 16
  Black or African-American | 2 | 4 | 6
  White | 123 | 111 | 234
  Other | 10 | 17 | 27
SF-36 Quality of life: Physical component summary [Mean (Standard Deviation); unit: units on a scale] — Short Form (36) Health Survey The SF-36 evaluates health-related quality of life in 8 domains consisting of two components: physical and mental. The score for each domain ranges from 0 to 100. Norm based scoring (based on the general US population) is used with a mean of 50 and standard deviation of 10. Higher values represent a better outcome.
  units on a scale | 45 (11) | 44 (11) | 44 (11)
SF-36 Quality of life: Mental component summary [Mean (Standard Deviation); unit: units on a scale] — Short Form (36) Health Survey The SF-36 evaluates health-related quality of life in 8 domains consisting of two components: physical and mental. The score for each domain ranges from 0 to 100. Norm based scoring (based on the general US population) is used with a mean of 50 and standard deviation of 10. Higher values represent a better outcome.
  units on a scale | 48 (12) | 48 (12) | 48 (12)
Liver enzymes: Alanine aminotransferase [Mean (Standard Deviation); unit: U/L] | 83 (49) | 82 (51) | 83 (50)
Liver enzymes: Aspartate aminotransferase [Mean (Standard Deviation); unit: U/L] | 64 (38) | 58 (34) | 61 (36)
Liver enzymes: Alkaline phosphatase [Mean (Standard Deviation); unit: U/L] | 82 (29) | 81 (25) | 82 (27)
Liver enzymes: γ-glutamyl transpeptidase [Mean (Standard Deviation); unit: U/L] | 78 (85) | 76 (97) | 77 (91)
Liver enzymes: Total bilirubin [Mean (Standard Deviation); unit: μmol/L] | 11.5 (5.9) | 11.3 (7.5) | 11.4 (6.8)
Lipids: Total cholesterol [Mean (Standard Deviation); unit: mmol/L] | 4.9 (1.2) | 4.8 (1.2) | 4.9 (1.2)
Lipids: HDL cholesterol [Mean (Standard Deviation); unit: mmol/L] | 1.1 (0.3) | 1.1 (0.4) | 1.1 (0.3)
Lipids: LDL cholesterol [Mean (Standard Deviation); unit: mmol/L] | 2.9 (1.0) | 2.9 (1.1) | 2.9 (1.0)
Lipids: Triglycerides [Mean (Standard Deviation); unit: mmol/L] | 2.2 (1.5) | 2.0 (1.7) | 2.1 (1.6)
Haematology: Haemoglobin [Mean (Standard Deviation); unit: g/L] | 140 (15) | 140 (14) | 140 (14)
Haematology: Haematocrit [Mean (Standard Deviation); unit: proportion of 1·0] | 0.41 (0.04) | 0.41 (0.04) | 0.41 (0.04)
Haematology: Mean corpuscular volume [Mean (Standard Deviation); unit: fL] | 88.7 (4.8) | 89.0 (5.3) | 88.9 (5.1)
Haematology: White blood cell count [Mean (Standard Deviation); unit: white blood cells *10^9 per L] | 7.3 (1.9) | 6.9 (2.3) | 7.1 (2.1)
Haematology: Platelet count [Mean (Standard Deviation); unit: platelets *10^9 per L] | 237 (59) | 237 (65) | 237 (62)
Chemistries: Bicarbonate [Mean (Standard Deviation); unit: mmol/L] | 25.9 (2.5) | 26.2 (2.6) | 26.0 (2.5)
Chemistries: Calcium [Mean (Standard Deviation); unit: mmol/L] | 2.4 (0.1) | 2.4 (0.1) | 2.4 (0.1)
Chemistries: Phosphate [Mean (Standard Deviation); unit: mmol/L] | 1.1 (0.2) | 1.1 (0.2) | 1.1 (0.2)
Chemistries: Creatinine [Mean (Standard Deviation); unit: μmol/L] | 71 (18) | 70 (16) | 71 (17)
Chemistries: Uric acid [Mean (Standard Deviation); unit: μmol/L] | 375 (89) | 366 (86) | 370 (87)
Chemistries: Albumin [Mean (Standard Deviation); unit: g/L] | 43 (4) | 43 (4) | 43 (4)
Chemistries: Total protein [Mean (Standard Deviation); unit: g/L] | 73 (5) | 74 (5) | 73 (5)
Other laboratory results: Prothrombin time [Mean (Standard Deviation); unit: s] | 11.7 (2.1) | 11.7 (2.2) | 11.7 (2.1)
Other laboratory results: International normalised ratio [Mean (Standard Deviation); unit: ratio] | 1.01 (0.08) | 1.00 (0.07) | 1.00 (0.07)
Metabolic factors: Fasting serum glucose [Mean (Standard Deviation); unit: mmol/L] | 6.5 (1.8) | 6.4 (2.2) | 6.4 (2.0)
Metabolic factors: Insulin [Mean (Standard Deviation); unit: pmol/L] | 201 (226) | 138 (129) | 169 (186)
Metabolic factors: HOMA-IR [Mean (Standard Deviation); unit: glucose [mmol/L] × insulin [pmol/L]/22.5] | 61 (74) | 40 (42) | 50 (61)
Metabolic factors: Glycated haemoglobin A1c [Mean (Standard Deviation); unit: mmol/mol] | 48 (12) | 47 (11) | 47 (11)
Metabolic factors: Weight [Mean (Standard Deviation); unit: kg] | 100 (23) | 96 (18) | 98 (21)
Metabolic factors: Body-mass index [Mean (Standard Deviation); unit: kg/m²] | 35 (7) | 34 (6) | 35 (6)
Metabolic factors: Waist circumference [Mean (Standard Deviation); unit: cm] | 112 (15) | 109 (14) | 111 (15)
Metabolic factors: Waist-to-hip ratio [Mean (Standard Deviation); unit: ratio] | 0.96 (0.07) | 0.95 (0.09) | 0.95 (0.08)
Metabolic factors: Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 132 (17) | 132 (15) | 132 (16)
Metabolic factors: Diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 77 (11) | 78 (10) | 77 (10)
Comorbidities: Hyperlipidaemia [Number; unit: participants] — History of cholesterol or triglyceride elevations as determined by the site investigator.
  participants | 87 | 86 | 173
Comorbidities: Hypertension [Number; unit: participants] | 87 | 85 | 172
Comorbidities: Cardiovascular disease [Number; unit: participants] | 7 | 8 | 15
Comorbidities: Diabetes [Number; unit: participants] | 75 | 74 | 149
Concomitant medications in the past 6 months: Antilipidaemic [Number; unit: participants] | 72 | 64 | 136
Concomitant medications in the past 6 months: Cardiovascular [Number; unit: participants] | 97 | 92 | 189
Concomitant medications in the past 6 months: Antidiabetic [Number; unit: participants] | 67 | 73 | 140
Concomitant medications in the past 6 months: Metformin [Number; unit: participants] | 55 | 62 | 117
Concomitant medications in the past 6 months: Pioglitazone [Number; unit: participants] | 1 | 6 | 7
Concomitant medications in the past 6 months: Vitamin E [Number; unit: participants] | 29 | 32 | 61
Concomitant medications in the past 6 months: Thiazolidinedione [Number; unit: participants] | 3 | 5 | 8
Concomitant medications in the past 6 months: Aspirin (81 mg) [Number; unit: participants] | 37 | 33 | 70
Liver histology findings: Definite steatohepatitis [Number; unit: participants] | 114 | 111 | 225
Liver histology findings: Fibrosis stage [Mean (Standard Deviation); unit: units on a scale] — †Fibrosis was assessed on a scale of 0-4, with higher scores showing more severe fibrosis.
  units on a scale | 1.9 (1.1) | 1.8 (1.0) | 1.8 (1.1)
Liver histology findings: Total NAFLD activity score [Mean (Standard Deviation); unit: units on a scale] — Total non-alcoholic fatty liver disease (NAFLD) activity was assessed on a scale of 0-8, with higher scores indicating more severe disease; the components of this measure are steatosis (assessed on a scale of 0-3), lobular inflammation (assessed on a scale of 0-3), and hepatocellular ballooning assessed on a scale of 0-2).
  units on a scale | 5.3 (1.3) | 5.1 (1.3) | 5.2 (1.3)
Liver histology findings: Hepatocellular ballooning score [Mean (Standard Deviation); unit: units on a scale] — Assessed on a scale of 0-2 with higher scores showing more severe ballooning.
  units on a scale | 1.4 (0.7) | 1.3 (0.7) | 1.4 (0.7)
Liver histology findings: Steatosis score [Mean (Standard Deviation); unit: units on a scale] — Assessed on a scale of 0-3 with higher scores showing more severe steatosis.
  units on a scale | 2.1 (0.8) | 2.0 (0.8) | 2.0 (0.8)
Liver histology findings: Lobular inflammation score [Mean (Standard Deviation); unit: units on a scale] — Assessed on a scale of 0-3 with higher scores showing more severe lobular inflammation.
  units on a scale | 1.8 (0.7) | 1.8 (0.7) | 1.8 (0.7)
Liver histology findings: Portal inflammation score [Mean (Standard Deviation); unit: units on a scale] — Portal inflammation was assessed on a scale of 0-2 with higher scores showing more severe inflammation.
  units on a scale | 1.2 (0.6) | 1.1 (0.6) | 1.1 (0.6)
Liver histology findings: Biopsy length [Mean (Standard Deviation); unit: mm] | 21 (10) | 21 (10) | 21 (10)

OUTCOME MEASURES:

1. Primary Outcome: Hepatic Histological Improvement in Nonalcoholic Fatty Liver Disease (NAFLD) Activity Score (NAS)
Description: Centrally scored histological improvement in nonalcoholic fatty liver disease (NAFLD) from baseline to the end of 72 weeks of treatment, where improvement is defined as:
  1. No worsening in fibrosis; and
  2. A decrease in NAFLD Activity Score (NAS) of at least 2 points
Time Frame: baseline to 72 weeks
Population: Number of randomly assigned patients with observed or expected week 72 visit before protocol modified on Jan 6, 2014, to eliminate week 72 biopsy. 11 patients in the placebo group and eight in the obeticholic acid group had missing histological data at week 72, and the results for these patients were imputed as a lack of improvement.
Measure: Number; unit: participants
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 110 | 109
participants | 50 | 23
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel; p values and relative benefit were calculated with the Cochran-Mantel-Haenszel chi-square test, stratified by clinic and diabetes status; Risk Ratio (RR) = 1.9, 95% CI 2-sided [1.3 to 2.8] — obeticholic acid vs placebo

2. Secondary Outcome: Resolution of NASH Diagnosis
Description: Resolution of definite nonalcoholic steatohepatitis. Resolution defined as either not NAFLD, or NAFLD but not non-alcoholic steatohepatitis on week 72 biopsy
Time Frame: baseline to 72 weeks
Population: Number of patients with biopsy specimens at baseline and 72 weeks
Measure: Number; unit: participants
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 102 | 98
participants | 22 | 13
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.08, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.5, 95% CI 2-sided [0.9 to 2.6] — obeticholic acid vs placebo

3. Secondary Outcome: Fibrosis: Patient With Improvement
Description: Patients with improvement in fibrosis score. Fibrosis was assessed on a scale of 0-4, with higher scores showing more severe fibrosis.
Time Frame: baseline to 72 weeks
Population: Number of patients with biopsy specimens at baseline and 72 weeks
Measure: Number; unit: participants
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 102 | 98
participants | 36 | 19
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.8, 95% CI 2-sided [1.1 to 2.7] — obeticholic acid vs placebo

4. Secondary Outcome: Fibrosis: Change in Score
Description: Change in fibrosis score. Fibrosis was assessed on a scale of 0-4, with higher scores showing more severe fibrosis.
Time Frame: baseline to 72 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 102 | 98
units on a scale | -0.2 (1.0) | 0.1 (0.9)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.01, ANCOVA; calculated using ANCOVA, regressing change from baseline to 72 weeks on treatment group and baseline value of the outcome; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.6 to -0.1] — obeticholic acid vs placebo

5. Secondary Outcome: Total NAFLD Activity Score: Change in Score
Description: NAFLD activity score was assessed on a scale of 0-8, with higher scores showing more severe disease (the components of this measure are steatosis [assessed on a scale of 0-3], lobular inflammation [assessed on a scale of 0-3], and hepatocellular ballooning [assessed on a scale of 0-2]).
Time Frame: baseline to 72 weeks
Population: Number of patients with biopsy specimens at baseline and 72 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 102 | 98
units on a scale | -1.7 (1.8) | -0.7 (1.8)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Net) = -0.9, 95% CI 2-sided [-1.3 to -0.5] — obeticholic acid vs placebo

6. Secondary Outcome: Hepatocellular Ballooning: Patients With Improvement
Description: Patients with improvement in hepatocellular ballooning score. Hepatocellular ballooning was assessed on a scale of 0-2, with higher scores showing more severe ballooning.
Time Frame: baseline to 72 weeks
Population: Number of patients with biopsy specimens at baseline and 72 weeks
Measure: Number; unit: participants
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 102 | 98
participants | 47 | 30
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.03, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.5, 95% CI 2-sided [1.0 to 2.1] — obeticholic acid vs placebo

7. Secondary Outcome: Hepatocellular Ballooning: Change in Score
Description: Change in hepatocellular ballooning score. Hepatocellular ballooning was assessed on a scale of 0-2, with higher scores showing more severe ballooning.
Time Frame: baseline to 72 weeks
Population: Number of patients with biopsy specimens at baseline and 72 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 102 | 98
units on a scale | -0.5 (0.9) | -0.2 (0.9)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.03, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.5 to 0.0] — obeticholic acid vs placebo

8. Secondary Outcome: Steatosis: Patients With Improvement
Description: Patients with improvement in steatosis score. Steatosis was assessed on a scale of 0-3, with higher scores showing more severe steatosis.
Time Frame: baseline to 72 weeks
Population: Number of patients with biopsy specimens at baseline and 72 weeks
Measure: Number; unit: participants
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 102 | 98
participants | 62 | 37
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.7, 95% CI 2-sided [1.2 to 2.3] — obeticholic acid vs. placebo

9. Secondary Outcome: Steatosis: Change in Score
Description: Change in steatosis score. Steatosis was assessed on a scale of 0-3, with higher scores showing more severe steatosis.
Time Frame: baseline to 72 weeks
Population: Number of patients with biopsy specimens at baseline and 72 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 102 | 98
units on a scale | -0.8 (1.0) | -0.4 (0.8)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.0004, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Net) = -0.4, 95% CI 2-sided [-0.6 to -0.2] — obeticholic acid vs placebo

10. Secondary Outcome: Lobular Inflammation: Patients With Improvement
Description: Patients with improvement in lobular inflammation score. Lobular inflammation was assessed on a scale of 0-3, with higher scores showing more severe lobular inflammation.
Time Frame: baseline to 72 weeks
Population: Number of patients with biopsy specimens at baseline and 72 weeks
Measure: Number; unit: participants
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 102 | 98
participants | 54 | 34
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.6, 95% CI 2-sided [1.1 to 2.2] — obeticholic acid vs. placebo

11. Secondary Outcome: Lobular Inflammation: Change in Score
Description: Change in lobular inflammation score. Lobular inflammation was assessed on a scale of 0-3, with higher scores showing more severe lobular inflammation.
Time Frame: baseline to 72 weeks
Population: Number of patients with biopsy specimens at baseline and 72 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 102 | 98
units on a scale | -0.5 (0.8) | -0.2 (0.9)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.0006, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.5 to -0.1] — obeticholic acid vs placebo

12. Secondary Outcome: Portal Inflammation: Patients With Improvement
Description: Patients with improvement in portal inflammation score. Portal inflammation was assessed on a scale of 0-2, with higher scores showing more severe portal inflammation.
Time Frame: baseline to 72 weeks
Population: Number of patients with biopsy specimens at baseline and 72 weeks
Measure: Number; unit: participants
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 102 | 98
participants | 12 | 13
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.90, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.0, 95% CI 2-sided [0.6 to 1.7] — obeticholic acid vs. placebo

13. Secondary Outcome: Portal Inflammation: Change in Score
Description: Change in portal inflammation score. Portal inflammation was assessed on a scale of 0-3, with higher scores showing more severe portal inflammation.
Time Frame: baseline to 72 weeks
Population: Number of patients with biopsy specimens at baseline and 72 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 102 | 98
units on a scale | 0.2 (0.7) | 0.2 (0.7)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.59, ANCOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.1 to 0.2] — obeticholic acid vs placebo

14. Secondary Outcome: Change in Alanine Aminotransferase
Time Frame: baseline to 72 weeks
Population: All patients who completed their final on-treatment study visit and the visit 24 weeks after stopping treatment (including those without a final biopsy due to early treatment termination) were included in the group comparisons of non-histological secondary outcomes.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
U/L | -38 (47) | -18 (44)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; calculated using ANCOVA models, regressing change from baseline to 72 weeks on treatment group and baseline value of the outcome; Mean Difference (Net) = -20, 95% CI 2-sided [-28 to -11] — obeticholic acid vs placebo

15. Secondary Outcome: Change in Asparate Aminotransferase
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
U/L | -27 (37) | -10 (31)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.0001, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = -12, 95% CI 2-sided [-18 to -6] — obeticholic acid vs placebo

16. Secondary Outcome: Change in Alkaline Phosphatase
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
U/L | 12 (26) | -6 (20)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = 18, 95% CI 2-sided [13 to 24] — obeticholic acid vs placebo

17. Secondary Outcome: Change in γ-glutamyl Transpeptidase
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
U/L | -37 (70) | -6 (48)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = -24, 95% CI 2-sided [-35 to -14] — obeticholic acid vs placebo

18. Secondary Outcome: Change in Total Bilirubin
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
μmol/L | -1.0 (4.1) | 0.6 (3.7)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = -1.5, 95% CI 2-sided [-2.4 to -0.5] — obeticholic acid vs placebo

19. Secondary Outcome: Change in Total Cholesterol
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
mmol/L | 0.16 (1.07) | -0.19 (0.96)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.0009, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = 0.38, 95% CI 2-sided [0.16 to 0.60] — obeticholic acid vs placebo

20. Secondary Outcome: Change in HDL Cholesterol
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
mmol/L | -0.02 (0.20) | 0.03 (0.19)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.01, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.10 to -0.01] — obeticholic acid vs placebo

21. Secondary Outcome: Change in LDL Cholesterol
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
mmol/L | 0.22 (0.90) | -0.22 (0.80)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = 0.45, 95% CI 2-sided [0.26 to 0.65] — obeticholic acid vs placebo

22. Secondary Outcome: Change in Triglycerides
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
mmol/L | -0.22 (1.27) | -0.08 (1.74)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.88, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.35 to 0.30] — obeticholic acid vs placebo

23. Secondary Outcome: Change in Haemoglobin
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
g/L | 0.6 (9.6) | 0.3 (9.5)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.72, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = 0.4, 95% CI 2-sided [-1.8 to 2.6] — obeticholic acid vs placebo

24. Secondary Outcome: Change in Haematocrit
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: proportion of 1.0
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
proportion of 1.0 | 0.00 (0.03) | 0.00 (0.03)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.71, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.01 to 0.01] — obeticholic acid vs placebo

25. Secondary Outcome: Change in Mean Corpuscular Volume
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
fL | -0.8 (2.6) | 0.3 (3.5)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = -1.1, 95% CI 2-sided [-1.8 to -0.4] — obeticholic acid vs placebo

26. Secondary Outcome: Change in White Blood Cell Count
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: white blood cells *10^9 per L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
white blood cells *10^9 per L | 0.0 (1.5) | 0.0 (1.1)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.40, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.2 to 0.4] — obeticholic acid vs placebo

27. Secondary Outcome: Change in Platelet Count
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: platelets *10^9 per L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
platelets *10^9 per L | 12 (33) | -4 (46)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = 16, 95% CI 2-sided [7 to 26] — obeticholic acid vs placebo

28. Secondary Outcome: Change in Bicarbonate
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
mmol/L | -0.7 (3.2) | -0.1 (2.7)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.03, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = -0.7, 95% CI 2-sided [-1.4 to -0.1] — obeticholic acid vs placebo

29. Secondary Outcome: Change in Calcium
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
mmol/L | 0.01 (0.10) | -0.01 (0.11)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.04, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = 0.02, 95% CI 2-sided [0.00 to 0.04] — obeticholic acid vs placebo

30. Secondary Outcome: Change in Phosphate
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
mmol/L | 0.01 (0.18) | 0.02 (0.16)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.53, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.03 to 0.05] — obeticholic acid vs placebo

31. Secondary Outcome: Change in Creatinine
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
μmol/L | 1.5 (11.3) | -1.1 (9.6)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.03, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = 2.6, 95% CI 2-sided [0.2 to 5.0] — obeticholic acid vs placebo

32. Secondary Outcome: Change in Uric Acid
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
μmol/L | 2 (68) | -11 (56)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.05, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = 14, 95% CI 2-sided [0 to 29] — obeticholic acid vs placebo

33. Secondary Outcome: Change in Albumin
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: gl/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
gl/L | -0.2 (3.1) | 0.3 (3.1)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.13, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.2 to 0.2] — obeticholic acid vs placebo

34. Secondary Outcome: Change in Total Protein
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: gl/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
gl/L | 0.2 (4.5) | -0.5 (4.5)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.31, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = 0.5, 95% CI 2-sided [-0.5 to 1.6] — obeticholic acid vs placebo

35. Secondary Outcome: Change in Prothrombin Time
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: s
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
s | -0.1 (2.4) | 0.0 (2.2)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.16, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.6 to 0.1] — obeticholic acid vs placebo

36. Secondary Outcome: Change in International Normalised Ratio
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
ratio | -0.03 (0.07) | 0.00 (0.08)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.04 to -0.01] — obeticholic acid vs placebo

37. Secondary Outcome: Change in Fasting Serum Glucose
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
mmol/L | 0.4 (2.1) | 0.2 (2.3)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.26, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.2 to 0.8] — obeticholic acid vs placebo

38. Secondary Outcome: Change in Insulin
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
pmol/L | 29 (159) | 10 (111)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.02, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = 38, 95% CI 2-sided [6 to 69] — obeticholic acid vs placebo

39. Secondary Outcome: Change in HOMA-IR
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: glucose[mmol/L]× insulin[pmol/L] / 22.5
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
glucose[mmol/L]× insulin[pmol/L] / 22.5 | 15 (50) | 4 (29)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.01, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = 13, 95% CI 2-sided [3 to 23] — obeticholic acid vs placebo

40. Secondary Outcome: Change in Glycated Haemoglobin A1c
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
mmol/mol | 0.5 (9.7) | 0.4 (8.3)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.71, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = 0.4, 95% CI 2-sided [-1.7 to 2.6] — obeticholic acid vs placebo

41. Secondary Outcome: Change in Weight
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
kg | -2.3 (6.7) | 0.0 (6.1)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.008, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = -2.2, 95% CI 2-sided [-3.7 to -0.6] — obeticholic acid vs placebo

42. Secondary Outcome: Change in Body-mass Index
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: kg/m²
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
kg/m² | -0.7 (2.4) | 0.1 (2.2)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.01, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = -0.7, 95% CI 2-sided [-1.3 to -0.2] — obeticholic acid vs placebo

43. Secondary Outcome: Change in Waist Circumference
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
cm | -1.5 (7.1) | -0.6 (8.7)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.70, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = -0.4, 95% CI 2-sided [-2.2 to 1.5] — obeticholic acid vs placebo

44. Secondary Outcome: Change in Waist-to-hip Ratio
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
ratio | 0.00 (0.06) | 0.00 (0.06)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.57, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = 0.00, 95% CI 2-sided [-0.01 to 0.02] — obeticholic acid vs placebo

45. Secondary Outcome: Change in Systolic Blood Pressure
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
mm Hg | -4 (17) | -1 (16)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.05, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = -3, 95% CI 2-sided [-7 to 0] — obeticholic acid vs placebo

46. Secondary Outcome: Change in Diastolic Blood Pressure
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
mm Hg | 0 (11) | 0 (10)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.23, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = -1, 95% CI 2-sided [-4 to 1] — obeticholic acid vs placebo

47. Secondary Outcome: Change in SF-36 Quality of Life Physical Component Summary
Description: Short Form (36) Health Survey The SF-36 evaluates health-related quality of life in 8 domains consisting of two components: physical and mental. The score for each domain ranges from 0 to 100. Norm based scoring (based on the general US population) is used with a mean of 50 and standard deviation of 10. Higher values represent a better outcome.
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
units on a scale | 0 (7) | -1 (7)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.22, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = 1, 95% CI 2-sided [-1 to 3] — obeticholic acid vs placebo

48. Secondary Outcome: Change in SF-36 Quality of Life Mental Component Summary
Description: as for outcome 47
Time Frame: baseline to 72 weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Obeticholic Acid | Placebo
Number analyzed (Participants) | 126 | 131
units on a scale | 0 (9) | 1 (9)
Statistical Analysis 1: Comparison: Obeticholic Acid vs Placebo; Test type: Superiority or Other; p = 0.65, ANCOVA; [statistical method as in outcome 14, analysis 1]; Mean Difference (Net) = 0, 95% CI 2-sided [-3 to 2] — obeticholic acid vs placebo

ADVERSE EVENTS:
Arm/Group | Obeticholic Acid | Placebo
Serious Adverse Events (participants affected / at risk) | 13/141 | 10/142
Other Adverse Events (participants affected / at risk) | 99/141 | 68/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obeticholic Acid (N=141) | Placebo (N=142)
Cardiovascular death or non-fatal myocardial infarction or non-fatal stroke (Cardiac disorders) | 3 (3) | 1 (2)
Other coronary artery disease or angina (Cardiac disorders) | 2 (2) | 2 (2)
Other cardiovascular event (Cardiac disorders) | 1 (1) | 1 (1)
Other neurological event (Nervous system disorders) | 1 (1) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hepatobiliary events (Hepatobiliary disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Other gastrointestinal event (Gastrointestinal disorders) | 2 (2) | 0 (0)
Other renal event (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obeticholic Acid (N=141) | Placebo (N=142)
Other cardiovascular event (Cardiac disorders) | 7 (7) | 5 (5)
Dizziness or syncope (Nervous system disorders) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 2 (2) | 5 (5)
Neuralgia (Nervous system disorders) | 3 (3) | 2 (2)
Other neurological event (Nervous system disorders) | 4 (4) | 8 (8)
Urinary tract infection or cystitis (Renal and urinary disorders) | 2 (2) | 3 (3)
Kidney stones (Renal and urinary disorders) | 6 (6) | 2 (2)
Other renal event (Renal and urinary disorders) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 32 (32) | 9 (9)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 7 (7)
Dental or tooth pain (Gastrointestinal disorders) | 4 (4) | 1 (1)
Liver pain post biopsy (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea, vomiting, or diarrhoea (Gastrointestinal disorders) | 12 (12) | 12 (12)
Constipation (Gastrointestinal disorders) | 5 (5) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Other gastrointestinal event (Gastrointestinal disorders) | 7 (7) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No